CLINICAL TRIAL: NCT00191815
Title: Phase II Study of Gemcitabine Plus Cisplatin as First-line Treatment of Metastatic Breast Cancer
Brief Title: Combination Chemotherapy for Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7311; B9E-VI-S326
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2009-08-19 (Estimated); Last update posted 2009-11-11 (Estimated); Status verified 2009-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gemcitabine; Cisplatin

ARMS (1):
- Gemcitabine + Cisplatin (Experimental)
  Interventions: Drug: Gemcitabine; Drug: cisplatin

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine (30 min intravenous infusion) dose of 1000mg/m2 on Day 1 and Day 8 (21 day cycle).
Drug: cisplatin — Cisplatin (30-120 min intravenous infusion) dose of 35 mg/m2 on Day 1 and Day 8 (21 day cycle).

SUMMARY:
The purpose of this study is to determine the objective tumor response of the first-line therapy combination of gemcitabine and cisplatin in patients with metastatic breast cancer

ELIGIBILITY:
Inclusion Criteria:

* You are female in the age of 18 to 75 years old.
* You have been diagnosed with the metastatic breast cancer.
* You have desire and an opportunity to visit your doctor in medical site, both during realization of the active treatment program, and within 24 months of medical follow up.
* You must sign this informed consent form

Exclusion Criteria:

* You are pregnant or breastfeeding.
* Your laboratory parameters fall outside the limits, admitted by requirements of the present clinical study.
* You have been diagnosed with serious concomitant or acute infectious disease.
* You have used experimental medications within the last month.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2002-10; Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5PM Eastern time (UTC/GMT - 5 hours, EST),, Study Director — Eli Lilly and Company
Locations (2):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon- Fri from 9AM to 5PM Eastern time (UTC/ GMT - 5hours, EST), or speak with your personal physician, Munich, Germany
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon- Fri from 9AM to 5PM Eastern time (UTC/ GMT - 5hours, EST), or speak with your personal physician, Moscow, Russia

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Gemcitabine + Cisplatin: Gemcitabine (30 min intravenous infusion) dose of 1000mg/m2 on Day 1 and Day 8 (21 day cycle).
  Cisplatin (30-120 min intravenous infusion) dose of 35 mg/m2 on Day 1 and Day 8 (21 day cycle).
Period: Overall Study
Arm/Group | Gemcitabine + Cisplatin
Started | 70
Treated | 67
Completed | 30
Not Completed | 40
Not completed — Adverse Event | 2
Not completed — Disease progression or relapse | 24
Not completed — Death | 2
Not completed — Protocol Violation | 3
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 7

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine + Cisplatin
Number analyzed (Participants) | 70
Age Continuous [Mean (Standard Deviation); unit: years] | 50.5 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 0
Region of Enrollment [Number; unit: participants]
  Russian Federation | 63
  Germany | 7
Menopausal Status [Number; unit: participants]
  Pre-menopausal | 16
  Post-menopausal | 54
Pathological Diagnosis [Number; unit: participants]
  Ductal breast carcinoma | 44
  Ductal and lobular breast carcinoma | 2
  Lobular breast carcinoma | 5
  Mucinous breast carcinoma | 1
  Adenocystic breast carcinoma | 10
  Papillary carcinoma | 1
  Unknown | 7
Stage of Disease at Entry to the Study [Number; unit: participants] — Stage of disease was determined using American Joint Committee on Cancer Staging Criteria for Breast Cancer. The higher the stage, the more severe the disease.
  participants
    Stage IIIb | 1
    Stage IV | 69
Stage of Disease at Time of Diagnosis [Number; unit: participants] — Stage of disease was determined using American Joint Committee on Cancer Staging Criteria for Breast Cancer. The higher the stage, the more severe the disease.
  participants
    Stage I | 3
    Stage IIa | 13
    Stage IIb | 22
    Stage IIIa | 12
    Stage IIIb | 15
    Stage IV | 5
Time from Initial Diagnosis to Study Entry [Mean (Standard Deviation); unit: month] | 37.6 (39.7)

OUTCOME MEASURES:

1. Primary Outcome: Objective Tumor Response
Description: Best response recorded from the start of treatment until disease progression/recurrence using World Health Organization (WHO) criteria that defines when participants improve ("respond"), stay the same ("stable"), or worsen ("progression") during treatment.
Time Frame: baseline to measured progressive disease (eight 21-day cycles of therapy and follow-up period was 24 months starting from the date of the last drug administration. Data collected every 4 months.)
Population: Efficacy Population: all enrolled participants who received study drug; did not have more than one neoadjuvant/adjuvant chemotherapy; had measurable disease; had prior neoadjuvant/adjuvant chemotherapy; and did not have prior chemotherapy for metastatic disease.
Measure: Number; unit: participants
Arm/Group | Gemcitabine + Cisplatin
Number analyzed (Participants) | 54
participants
  Complete Response | 7
  Partial Response | 19
  Stable Disease | 19
  Progressive Disease | 5
  Not Assessable | 4

2. Secondary Outcome: Duration of Response
Description: The duration of a complete response (CR) or partial response (PR) was defined as the time from first objective status assessment of CR or PR to the first time of progression or death as a result of any cause.
Time Frame: first documented complete or partial response to measured progressive disease (eight 21-day cycles of therapy and follow-up period was 24 months starting from the date of the last drug administration.)
Population: Response population: all enrolled participants who had either a complete or partial response.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Gemcitabine + Cisplatin
Number analyzed (Participants) | 26
weeks | 32.7 [26.9 to 48.6]

3. Secondary Outcome: Time to Progressive Disease
Description: Defined as the time from study enrollment to the first date of disease progression.
Time Frame: first active treatment dose to measured progressive disease (eight 21-day cycles of therapy and follow-up period was 24 months starting from the date of the last drug administration.)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Gemcitabine + Cisplatin
Number analyzed (Participants) | 54
weeks | 33.9 [23.9 to 48.0]

4. Secondary Outcome: Time to Treatment Failure
Description: Defined as the time from study enrollment to the first observation of disease progression, death as a result of any cause, or early discontinuation of treatment.
Time Frame: first active treatment dose to last contact for patients, death as a result of any cause, or early discontinuation of treatment (eight 21-day cycles of therapy and follow-up period was 24 months starting from the date of the last drug administration.)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Gemcitabine + Cisplatin
Number analyzed (Participants) | 54
weeks | 26.2 [19.6 to 34.9]

5. Secondary Outcome: Survival Time
Description: Overall survival is the duration from enrollment to death due to any cause.
Time Frame: first active treatment dose to date of death due to any cause (eight 21-day cycles of therapy and follow-up period was 24 months starting from the date of the last drug administration.)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Gemcitabine + Cisplatin
Number analyzed (Participants) | 54
weeks | 84.0 [58.6 to 119.3]

6. Secondary Outcome: Number of Participants With Maximum Common Toxicity Criteria-National Cancer Institute Toxicity (CTC-NCI) of Gemcitabine-Cisplatin Combination
Description: The CTC provides descriptive terminology for adverse event reporting. A grading (severity) scale is provided for each adverse event term. Grades range from 0 (none) to 5 (death).
Time Frame: Baseline up to 30 days after last dose of study drug (eight 21-day cycles of therapy)
Population: Safety Population: all enrolled participants who received study drug.
Measure: Number; unit: participants
Arm/Group | Gemcitabine + Cisplatin
Number analyzed (Participants) | 67
participants
  Allergic reaction/hypersensivity - Grade 1 | 1
  Allergic reaction/hypersensivity - Grade 2 | 1
  Allergic reaction/hypersensivity - Grade 3 | 0
  Allergic reaction/hypersensivity - Grade 4 | 0
  Allergic rhinitis - Grade 1 | 1
  Allergic rhinitis - Grade 2 | 0
  Allergic rhinitis - Grade 3 | 0
  Allergic rhinitis - Grade 4 | 0
  Other auditory/hearing - Grade 1 | 0
  Other auditory/hearing - Grade 2 | 0
  Other auditory/hearing - Grade 3 | 1
  Other auditory/hearing - Grade 4 | 0
  Blood/Bone marrow - other - Grade 1 | 0
  Blood/Bone marrow - other - Grade 2 | 0
  Blood/Bone marrow - other - Grade 3 | 0
  Blood/Bone marrow - other - Grade 4 | 1
  Cardiac- ischemia/infarction - Grade 1 | 0
  Cardiac- ischemia/infarction - Grade 2 | 0
  Cardiac- ischemia/infarction - Grade 3 | 1
  Cardiac- ischemia/infarction - Grade 4 | 0
  Hypertension - Grade 1 | 0
  Hypertension - Grade 2 | 1
  Hypertension - Grade 3 | 0
  Hypertension - Grade 4 | 0
  Hypotension - Grade 1 | 0
  Hypotension - Grade 2 | 0
  Hypotension - Grade 3 | 0
  Hypotension - Grade 4 | 1
  Fatigue - Grade 1 | 6
  Fatigue - Grade 2 | 1
  Fatigue - Grade 3 | 0
  Fatigue - Grade 4 | 0
  Fever - Grade 1 | 0
  Fever - Grade 2 | 1
  Fever - Grade 3 | 0
  Fever - Grade 4 | 0
  Rigors, chills - Grade 1 | 1
  Rigors, chills - Grade 2 | 0
  Rigors, chills - Grade 3 | 0
  Rigors, chills - Grade 4 | 0
  Weight loss - Grade 1 | 1
  Weight loss - Grade 2 | 1
  Weight loss - Grade 3 | 0
  Weight loss - Grade 4 | 0
  Alopecia - Grade 1 | 1
  Alopecia - Grade 2 | 3
  Alopecia - Grade 3 | 0
  Alopecia - Grade 4 | 0
  Rash/desquamation - Grade 1 | 0
  Rash/desquamation - Grade 2 | 0
  Rash/desquamation - Grade 3 | 1
  Rash/desquamation - Grade 4 | 0
  Anorexia - Grade 1 | 4
  Anorexia - Grade 2 | 0
  Anorexia - Grade 3 | 0
  Anorexia - Grade 4 | 0
  Constipation - Grade 1 | 1
  Constipation - Grade 2 | 0
  Constipation - Grade 3 | 0
  Constipation - Grade 4 | 0
  Mucositis due to radiation - Grade 1 | 2
  Mucositis due to radiation - Grade 2 | 0
  Mucositis due to radiation - Grade 3 | 0
  Mucositis due to radiation - Grade 4 | 0
  Nausea - Grade 1 | 10
  Nausea - Grade 2 | 8
  Nausea - Grade 3 | 2
  Nausea - Grade 4 | 0
  Vomiting - Grade 1 | 4
  Vomiting - Grade 2 | 7
  Vomiting - Grade 3 | 1
  Vomiting - Grade 4 | 0
  SGPT (ALT) - Grade 1 | 0
  SGPT (ALT) - Grade 2 | 1
  SGPT (ALT) - Grade 3 | 0
  SGPT (ALT) - Grade 4 | 0
  Infection without neutropenia - Grade 1 | 1
  Infection without neutropenia - Grade 2 | 0
  Infection without neutropenia - Grade 3 | 0
  Infection without neutropenia - Grade 4 | 0
  Insomnia - Grade 1 | 0
  Insomnia - Grade 2 | 0
  Insomnia - Grade 3 | 1
  Insomnia - Grade 4 | 0
  Abdominal pain or cramping - Grade 1 | 1
  Abdominal pain or cramping - Grade 2 | 1
  Abdominal pain or cramping - Grade 3 | 0
  Abdominal pain or cramping - Grade 4 | 0
  Headache - Grade 1 | 0
  Headache - Grade 2 | 0
  Headache - Grade 3 | 1
  Headache - Grade 4 | 0
  Pain - Other - Grade 1 | 0
  Pain - Other - Grade 2 | 0
  Pain - Other - Grade 3 | 1
  Pain - Other - Grade 4 | 0
  Renal/Genitourinary - Other - Grade 1 | 1
  Renal/Genitourinary - Other - Grade 2 | 0
  Renal/Genitourinary - Other - Grade 3 | 1
  Renal/Genitourinary - Other - Grade 4 | 0

7. Secondary Outcome: Number of Participants With Hematology Maximum Common Toxicity Criteria - National Cancer Institute Grades
Description: Maximum CTC-NCI toxicity grade for hematology. Grades range from 0 (none) to 5 (death).
Time Frame: Baseline up to 30 days after last dose of study drug (eight 21-day cycles of therapy)
Population: Safety Population: all enrolled participants who received study drug.
Measure: Number; unit: participants
Arm/Group | Gemcitabine + Cisplatin
Number analyzed (Participants) | 67
participants
  Hemoglobin (g/L) - Grade 1 | 35
  Hemoglobin (g/L) - Grade 2 | 20
  Hemoglobin (g/L) - Grade 3 | 5
  Hemoglobin (g/L) - Grade 4 | 1
  Neutrophils (x10E9/L) - Grade 1 | 6
  Neutrophils (x10E9/L) - Grade 2 | 25
  Neutrophils (x10E9/L) - Grade 3 | 13
  Neutrophils (x10E9/L) - Grade 4 | 10
  Platelets (x10E9/L) - Grade 1 | 43
  Platelets (x10E9/L) - Grade 2 | 2
  Platelets (x10E9/L) - Grade 3 | 1
  Platelets (x10E9/L) - Grade 4 | 0
  White Blood Cells (x10E9/L) - Grade 1 | 16
  White Blood Cells (x10E9/L) - Grade 2 | 27
  White Blood Cells (x10E9/L) - Grade 3 | 18
  White Blood Cells (x10E9/L) - Grade 4 | 3

8. Secondary Outcome: Number of Deaths
Time Frame: Baseline through follow-up (eight 21-day cycles of therapy and follow-up period was 24 months starting from the date of the last drug administration.)
Population: All enrolled participants.
Measure: Number; unit: participants
Arm/Group | Gemcitabine + Cisplatin
Number analyzed (Participants) | 70
participants
  Disease Progression | 35
  Ventricular Fibrillation | 1
  Circulatory Arrest | 1

9. Secondary Outcome: Number of Participants With Adverse Events Leading to Discontinuation
Time Frame: Baseline through eight 21-day cycles
Population: Safety Population: all enrolled participants who received study drug.
Measure: Number; unit: participants
Arm/Group | Gemcitabine + Cisplatin
Number analyzed (Participants) | 67
participants
  Patients with >=1 AE leading to discontinuation | 2
  Pneumonia | 1
  Toxic skin eruption | 1

ADVERSE EVENTS:
Arm/Group | Gemcitabine + Cisplatin
Serious Adverse Events (participants affected / at risk) | 6
Other Adverse Events (participants affected / at risk) | 54
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Gemcitabine + Cisplatin
Atrial fibrillation (Cardiac disorders) | 1/67 (1)
Ventricular fibrillation (Cardiac disorders) | 1/67 (1)
Gastrointestinal perforation (Gastrointestinal disorders) | 1/67 (1)
Periproctitis (Gastrointestinal disorders) | 1/67 (1)
General physical health deterioration (General disorders) | 1/67 (1)
Escherichia sepsis (Infections and infestations) | 1/67 (1)
Pneumonia (Infections and infestations) | 1/67 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/67 (1)
Renal failure acute (Renal and urinary disorders) | 1/67 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1/67 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1/67 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1/67 (1)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1/67 (1)
Circulatory collapse (Vascular disorders) | 1/67 (1)
Thrombosis (Vascular disorders) | 1/67 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Gemcitabine + Cisplatin
Neutropenia (Blood and lymphatic system disorders) | 16/67 (26)
Nausea (Gastrointestinal disorders) | 23/67 (46)
Vomiting (Gastrointestinal disorders) | 12/67 (20)
Asthenia (General disorders) | 14/67 (29)
Weight decreased (Investigations) | 7/67 (7)
Hypercalcaemia (Metabolism and nutrition disorders) | 5/67 (6)
Hyperkalaemia (Metabolism and nutrition disorders) | 9/67 (12)
Hypocalcaemia (Metabolism and nutrition disorders) | 6/67 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 5/67 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 4/67 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days